CLINICAL TRIAL: NCT02175342
Title: Pharmacodynamic and Pharmacokinetic Dose Ranging Study of Tiotropium Bromide Administered Via Respimat Device in Patients With Chronic Obstructive Pulmonary Disease (COPD): a Randomized, 3-week Multiple-dose, Placebo Controlled, Intraformulation Double-blind, Parallel Group Study
Brief Title: Pharmacodynamic and Pharmacokinetic Dose Ranging Study of Tiotropium Bromide Administered Via Respimat Device in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.127
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (8):
- Tiotropium-1.25 Respimat (Experimental): Two puffs of tiotropium inhalation solution from a Respimat device, 0.625 mcg/puff
  Interventions: Drug: Tiotropium 0.625 mcg/puff; Device: Respimat
- Tiotropium-2.5 Respimat (Experimental): Two puffs of tiotropium inhalation solution from a Respimat device, 1.25 mcg/puff
  Interventions: Drug: Tiotropium 1.25 mcg/puff; Device: Respimat
- Tiotropium-5 Respimat (Experimental): Two puffs of tiotropium inhalation solution from a Respimat device, 2.5 mcg/puff
  Interventions: Drug: Tiotropium 2.5 mcg/puff; Device: Respimat
- Tiotropium-10 Respimat (Experimental): Two puffs of tiotropium inhalation solution from a Respimat device, 5 mcg/puff
  Interventions: Drug: Tiotropium 5 mcg/puff; Device: Respimat
- Tiotropium-20 Respimat (Experimental): Two puffs of tiotropium inhalation solution from a Respimat device, 10 mcg/puff
  Interventions: Drug: Tiotropium 10 mcg/puff; Device: Respimat
- Placebo Respimat (Placebo Comparator)
  Interventions: Drug: Placebo solution; Device: Respimat
- Tiotropium-18 lactose powder Handihaler (Active Comparator)
  Interventions: Drug: Tiotropium-18 lactose powder; Device: Handihaler
- Placebo lactose powder Handihaler (Placebo Comparator)
  Interventions: Drug: Placebo lactose powder; Device: Handihaler

INTERVENTIONS:
Drug: Tiotropium 0.625 mcg/puff
  Arms: Tiotropium-1.25 Respimat
Drug: Tiotropium 1.25 mcg/puff
  Arms: Tiotropium-2.5 Respimat
Drug: Tiotropium 2.5 mcg/puff
  Arms: Tiotropium-5 Respimat
Drug: Tiotropium 5 mcg/puff
  Arms: Tiotropium-10 Respimat
Drug: Placebo solution
  Arms: Placebo Respimat
Drug: Tiotropium-18 lactose powder
  Arms: Tiotropium-18 lactose powder Handihaler
Drug: Placebo lactose powder
  Arms: Placebo lactose powder Handihaler
Drug: Tiotropium 10 mcg/puff
  Arms: Tiotropium-20 Respimat
Device: Respimat
  Arms: Placebo Respimat; Tiotropium-1.25 Respimat; Tiotropium-10 Respimat; Tiotropium-2.5 Respimat; Tiotropium-20 Respimat; Tiotropium-5 Respimat
Device: Handihaler
  Arms: Placebo lactose powder Handihaler; Tiotropium-18 lactose powder Handihaler

SUMMARY:
This pharmacodynamic and pharmacokinetic dose-ranging study aims to determine the optimal dose of tiotropium inhaled as a solution from a Respimat device once a day for three weeks in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 40 years;
2. Diagnosis of COPD and met the following criteria:

   1. Relatively stable, moderate to severe airway obstruction,
   2. Baseline 30% ≤ FEV1 ≤ 65% of predicted normal value, predicted normal values are based on the guidelines for standardized lung function testing of the European Community for Coal and Steel (ECCS) ,
   3. Baseline FEV1/ forced expiratory vital capacity (FEVC) ≤ 70%;
3. Smoking history ≥ 10 pack-years (p.y.). A p.y. is defined as the equivalent of smoking one pack of cigarettes per day for one year;
4. Male of female;
5. Ability to be trained in the proper use of Respimat and Handihaler;
6. Ability to be trained in the performance of technically satisfactory pulmonary function tests;
7. Ability to provide written informed consent
8. Patient affiliated to the Social Security System

Exclusion Criteria:

1. History of asthma, allergic rhinitis or atopy or who have a blood eosinophil count above 600/mm³
2. Changes in the therapeutic (pulmonary) plan within the last six weeks prior to the Screening Visit;
3. Treatment by cromolyn/nedocromil sodium;
4. Treatment by antihistamines (H1 receptor antagonists);
5. A lower respiratory tract infection or any exacerbation in the past six weeks prior to the Screening Visit;
6. Regular use of daytime oxygen therapy;
7. Treatment by oral corticosteroid medication if initiated or modified within the last six weeks or if daily dose > 10 mg prednisone equivalent;
8. History of life threatening pulmonary obstruction, cystic fibrosis or bronchiectasis
9. Patients who have undergone thoracotomy with pulmonary resection;
10. History of clinically significant cardiovascular, renal neurologic, liver or endocrine dysfunction. A clinically significant disease was defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
11. Patients with a recent (≤ one year) history of myocardial infarction, of heart failure or patients with any cardiac arrhythmia requiring drug therapy;
12. Tuberculosis with indication for treatment;
13. History of cancer within the last five years. Patients with treated basal cell carcinoma were allowed:
14. Current psychiatric disorders;
15. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction;
16. Patients with any history of glaucoma or increased intra-ocular pressure;
17. Patients with clinically significant abnormal baseline haematology or blood chemistry, if the abnormality defines a disease listed as an exclusion criterion;
18. Patients with

    1. glutamyl-oxalo-acetic transaminase/glutamyl-pyruvic transaminase (SGOT/SGPT): > 200% of the upper limit of the normal range (ULN, )
    2. bilirubin: > 150% of the ULN,
    3. creatinine: > 125% of the ULN;
19. Intolerance to aerosolised anticholinergic containing products, and/or hypersensitivity to benzalkonium chloride, to lactose or any other components of the inhalation capsule delivery system;
20. Beta-blocker medication;
21. Concomitant or recent (within the last month) use of investigational drugs;
22. History of drug abuse and/or alcoholism;
23. Pregnant or nursing women and women of childbearing potential not using a medically approved means of contraception ( urinary pregnancy test at screening);
24. Previous participation in this study (i.e. having been allocated a randomised treatment number);
25. Patients deprived of their freedom by a judicial or administrative decision;
26. Minors, adults under guardianship;
27. Persons in medical or social establishments;
28. Patients in emergency situations

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 1998-03-01 (Actual); Primary Completion 1999-04-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) with emphasis on the last two hours of the 24-hour dosing interval (trough FEV1) | last two hours of the 24-hour dosing interval

SECONDARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | during the first four hours post dose
Forced Vital Capacity (FVC) | during first four hours post dose
Pharmacokinetic evaluation: 2-hours urine sampling pre- and post-dose (10 patients per group) | before and after last drug administration at day7,14 and 21.
Chronic obstructive pulmonary disease symptom scores, physician's global evaluation, sleep question and use of rescue medication | 3 weeks treatment period
Changes in ECG, pulse rate (PR) and blood pressure (BP) from the pre-dose values recorded on test day | Day 0, day 7, day 14, day 21
Changes in ECG, physical examination, haematology and biochemistry recorded before and after the trial | Screening, 24 to 28 days after treatment
Occurrence of adverse events | up to 28 days

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency